CLINICAL TRIAL: NCT00598052
Title: Treatment of Marijuana Withdrawal Syndrome Using Escitalopram and Cognitive-Behavior Therapy- a Double-Blind Placebo-Controlled Study
Brief Title: Treatment of Marijuana Withdrawal Syndrome Using Escitalopram and Cognitive-Behavior Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Miki Bloch, Sourasky Medical center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-7.1.08-CTIL; Sponsored by IADA
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-01

CONDITIONS: Marijuana Dependence
Keywords: Marijuana dependence withdrawal Escitalopram
MeSH Terms: conditions — Marijuana Abuse | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Escitalopram + cognitive-behavior treatment
  Interventions: Drug: Escitalopram
- B (Placebo Comparator): Placebo + cognitive-behavior therapy
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 10mg/day
  Other Names: Cipralex

SUMMARY:
Recent studies have established the reliability, validity and time course of the cannabis withdrawal syndrome. This study will investigate the effects of combined treatment of Escitalopram with cognitive-behavior therapy in alleviating the symptoms of the marijuana withdrawal syndrome in regular chronic users of marijuana. We predict that combined pharmacological treatment and cognitive-behavior therapy will help patients to abstain from using using marijuana and it will alleviate their marijuana withdrawal symptoms.

DETAILED DESCRIPTION:
Recent studies have established the reliability, validity and time course of the cannabis withdrawal syndrome characterized by symptoms of anxiety, irritability, negative mood, physical symptoms and decreased appetite. This study will investigate the effects of combined treatment of Escitalopram with cognitive-behavior therapy in alleviating the symptoms of the marijuana withdrawal syndrome in regular chronic users of marijuana. 40 patients will be blindly randomized to either active or placebo escitalopram 10mg/day, for 12 weeks followed bt 12 weeks of follow-up.

Inclusion criteria include:

* Men and women age 20-45
* DSM-IV diagnosis of THC dependence.

Exclusion criteria include:

* Dependence on other drugs or alcohol
* Bipolar Disorder or Schizophrenia, Major depression, suicidal ideation psychotic symptoms or violent thoughts
* Current treatment with anti-depressant medication
* Neurological disease
* Physical illness (hypothyroidism, severe anemia, renal failure)
* Past severe effects of SSRIs.

Outcome measures include:

* urine THC analysis every two weeks
* questionnaires assessing addiction severity index
* depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 20-45
* DSM IV criteria of marijuana dependence.

Exclusion Criteria:

* Other drug or alcohol dependence
* Bipolar disorder, schizophrenia, major depression, suicidal ideation, psychotic symptoms or violent thoughts
* Physical illness including hypothyroidism, neurological disease, severe anemia, and renal failure
* Past severe side effects of SSRIs.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Clean urine THC samples | Every 2 weeks

SECONDARY OUTCOMES:
Questionnaire ratings of anxiety and depression and withdrawal symptoms | Every week of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Miki Bloch, M.D, Principal Investigator — Sourasky Medical center, Tel Aviv; Aviv M Weinstein, Ph.D, Principal Investigator — Sourasky Medical Center Tel Aviv, Israel
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel